CLINICAL TRIAL: NCT05409326
Title: A Phase I Study of TQH2722 Injection to Evaluate the Safety, Tolerability, Pharmacokinetics, Efficacy and Immunogenicity in Healthy Adult Subjects
Brief Title: A Study of TQH2722 Injection to Evaluate the Safety, Tolerability, Pharmacokinetics, Efficacy and Immunogenicity in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2722-I-01
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH2722 injection (Experimental): Participants will receive single dose of TQH2722 injection under fasted condition (Single Ascending Dose(SAD) Cohorts 50mg, 150mg, 300mg, 600mg, 1200mg) on Day 1, or will receive multiple doses of TQH2722 injection once every 14 days under fasted condition (Multiple-Dose Administration (MAD) Cohort 150mg, 600mg) on Day 1-43.
  Interventions: Drug: TQH2722 injection
- Placebo to match TQH2722 (Placebo Comparator): Participants will receive single dose of matching placebo under fasted condition (Single Ascending Dose(SAD) Cohorts 50mg, 150mg, 300mg, 600mg, 1200mg) on Day 1, or will receive multiple doses of matching placebo once every 14 days under fasted condition (Multiple-Dose Administration (MAD) Cohort 150mg, 600mg) on Day 1-43.
  Interventions: Drug: Placebo to match TQH2722

INTERVENTIONS:
Drug: TQH2722 injection — TQH2722 is a fully human monoclonal antibody directed against the interleukin (IL)-4 receptor α subunit (IL-4Rα) of IL-4 heterodimeric type I and type II receptors that mediate IL-4/IL-13 signaling through this pathway. Blockade of these receptors broadly suppresses type 2 inflammation associated with atopic/allergic diseases.
  Arms: TQH2722 injection
Drug: Placebo to match TQH2722 — TQH2722 is a fully human monoclonal antibody directed against the interleukin (IL)-4 receptor α subunit (IL-4Rα) of IL-4 heterodimeric type I and type II receptors that mediate IL-4/IL-13 signaling through this pathway. Blockade of these receptors broadly suppresses type 2 inflammation associated with atopic/allergic diseases.
  Arms: Placebo to match TQH2722

SUMMARY:
A randomized, double-blind, placebo-controlled trial design was used to assess the safety, tolerability, pharmacokinetics and pharmacodynamics characteristics, and immunogenicity of TQH2722 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1 The informed consent was signed before the trial, fully understood the purpose and process of the trial and the possible adverse reactions.
* 2 Aged 18 ~ 60 years old (including the critical value), both male and female;
* 3 ≥ 45 kg for females and ≥ 50 kg for males with a body mass index (BMI) between 19 and 26 kg/m2 inclusive, BMI = weight (kg)/height2 (m2)
* 4 The subject is able to communicate well with the investigator, voluntary and able to understand and follow protocol procedures to complete the study;
* 5 The subject agrees not to have a childbearing plan from the date of signing the informed consent form to 6 months after the last dose, and must use effective non-drug contraception with a partner of childbearing potential;
* 6 Normal physical examination, vital signs or abnormal physical examination, vital signs without clinical significance

Exclusion Criteria:

* 1 Females who are pregnant, lactating or have unprotected sex within two weeks prior to screening;
* 2 Past medical history or current cardiac, endocrine, metabolic, renal, hepatic, gastrointestinal, skin, infection, hematological, neurological or psychiatric diseases/abnormalities, or related chronic diseases, or acute diseases, and the investigator evaluated that the subject was not suitable for the trial;
* 3 People who have abnormal and clinically significant results in vital signs, physical examination, laboratory tests, eye examination, 12-lead ECG and X-ray during screening period;
* 4 Subjects Positive for Any of Hepatitis B Virus Surface Antigen (HBsAg), Hepatitis C Virus Antibody (Anti-HCV), Human Immunodeficiency Virus Antibody (Anti-HIV), and Treponema Pallidum Antibody (Anti-TP);
* 5 Clinically significant respiratory infection requiring antibiotic or antiviral therapy within 7 days prior to randomization;
* 6 People who received surgical operation within 4 weeks prior to screening, or planned to receive surgical operation during the study period;
* 7 People who participated in other clinical trials and took the study drug within 3 months before screening;
* 8 Received immunoglobulins or blood products within 30 days prior to randomization;
* 9 Blood loss or blood donation of more than 400 mL within 2 months prior to randomization;
* 10 People who have potential difficulty in blood collection, or have a history of halo needles or blood sickness;
* 11 A history of allergic reactions to another therapeutic monoclonal antibody or biologic agent therapy, or any clear history of drug or food allergies, particularly those with allergies to similar components to the drug in this trial;
* 12 People who have received or are planning to receive live-reduced or active vaccines during the 30 days prior to randomization and the entire study period (including the follow-up period);
* 13 Smoking more than 5 cigarettes per day or using equivalent amounts of nicotine or nicotine-containing products during the 6 months prior to randomization and the entire study period (including the follow-up period);
* 14 People who had long-standing alcohol abuse or alcohol consumption of more than 14 units (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) of alcohol per week during the 3 months prior to screening and the entire study period (including the follow-up period), or those who tested positive for alcohol breath;
* 15 People with a history of substance abuse or positive urine drug screening;
* 16 Received any marketed or research biologics within 4 months or 5 half-lives (whichever is longer) prior to randomization;
* 17 Taking any prescription, over-the-counter and herbal medicines within 4 weeks prior to randomization, with the exception of vitamin products;
* 18 Use of any systemic cytotoxicity or systemic immunosuppressants within 6 months prior to randomization or during the study period, or any local cytotoxin or local immunosuppressive drug within 30 days or 5 half-life periods (whichever is longer) prior to randomization or during the study period;
* 19 Parasitic infection is associated and is excluded if any of the following are met:

  * During the screening period, the stool routinely checks positive for eggs;
  * History of parasitic infection within 6 months prior to the screening period;
  * Have traveled or planned to travel to endemic parasitic infection areas (including but not limited to Southeast and South-West Asia, South America and Africa) within 6 months prior to screening visits;
* 20 Any situation in which the investigator believes that this poses a safety risk to the subject in the trial or may interfere with the conduct of the study, or that the investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Incidence and severity of adverse events (AE) .
Serious adverse events (SAE) | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Incidence and severity of Serious adverse events (SAE).
Blood biochemistry | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal indicators of blood biochemistry.
Coagulation function | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal indicators of coagulation function.
Blood routine | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal indicators of blood routine.
Urinalysis | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal indicators of urinalysis.
Blood pressure | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal values of blood pressure
Pulse | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal values of blood pulse.
Body temperature | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal values of blood body temperature.
Skin | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the skin.
Mucous membranes | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the mucous membranes.
Lymph nodes | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the lymph nodes.
Head | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the head.
Neck | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the neck.
Chest | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the chest.
Abdomen | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the abdomen.
Spine | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the spine.
Limbs | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Examination of the limbs.
12-lead electrocardiogram | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 99 days.
  Abnormal values of 12-lead electrocardiogram

SECONDARY OUTCOMES:
Maximum Concentration（Cmax） | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Maximum Concentration
Minimum Concentration(Cmax) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Minimum Concentration
Time to maximum concentration(Tmax) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Time to maximum concentration following drug administration
Area under the drug-time curve(AUC) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Area under the drug-time curve
Apparent terminal elimination half-life(t1/2) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Apparent terminal elimination half-life following drug administration
Apparent volume of distribution(Vd/F) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose.
  Apparent volume of distribution
Clearance rate(CL/F) | SAD:Before administration,1,4,8,12,24,72,168,240,336,408,504,576,672,840,1008,1176,1344 hours postdose. MAD:Before every administration,1,4,8,12,24,72,168,504,840,1009,1012,1016,1020,1032,1080,1176,1334,1512,1680,1848,2016,2352 hours postdose
  Clearance rate
Immunoglobulin E(IgE) | SAD:Before administration,168,336,504,672,1008,1344 hours after administration. MAD:Before every administration,336,672,1344 hours after the last administration.
  Percentage of changes in serum IgE
Thymus activation regulates chemokines(TARC) | SAD:Before administration,168,336,504,672,1008,1344 hours after administration. MAD:Before every administration,336,672,1344 hours after the last administration.
  Percentage of changes in serum TARC
Anti-drug antibody (ADA) | SAD:Before administration,336,1344 hours after administration. MAD:Before the first administration;Before the third administration;336,1344 hours after the last administration.
  Incidence and titer of anti-drug antibody
Neutralizing Antibody(Nab) | SAD:Before administration,336,1344 hours after administration. MAD:Before the first administration;Before the third administration;336,1344 hours after the last administration.
  Incidence of Neutralizing Antibody
Injection site response | Before administration,0.5,1,3,6 hours after administration.
  Injection site response assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China